CLINICAL TRIAL: NCT06251258
Title: Facial Emotion Recognition in Insomnia and Emotional Regulation
Acronym: REFIRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-A02559-36
Record Dates: First submitted 2024-01-16; First posted 2024-02-09 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Chronic Insomnia
Keywords: chronic insomnia; neuropsychology; facial expression assessment; emotional regulation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Emotional Regulation | interventions — Eye-Tracking Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insomnia (Experimental)
  Interventions: Diagnostic Test: Facial emotion recognition test with and without eye-tracking and Cognitive Emotion Regulation. Questionnaire (CERQ)
- Control (Active Comparator)
  Interventions: Diagnostic Test: Facial emotion recognition test with and without eye-tracking and Cognitive Emotion Regulation. Questionnaire (CERQ)

INTERVENTIONS:
Diagnostic Test: Facial emotion recognition test with and without eye-tracking and Cognitive Emotion Regulation. Questionnaire (CERQ) — Facial emotion recognition test without eye-tracking (explicit test, without time limit) and facial emotion recognition test with eye tracking (implicit test, with observation of fixation points)

SUMMARY:
Introduction Chronic insomnia is a prevalent disorder in the general population, affecting up to 20% according to French National Institute of Health and Medical Research, leading to a decline in quality of life and an increased risk of developing certain psychiatric disorders, notably major depressive episodes. Chronic insomnia, particularly when accompanied by reduced sleep duration, has been associated with cognitive impairments documented in the literature, such as reduced concentration, working memory, vigilance, and certain executive functions.

While some studies suggest subjective cognitive impairment in insomnia, it remains inconclusive when objectively measured. Individuals with chronic insomnia often report a global deterioration in social life, characterized by irritability, attentional difficulties, asthenia, and social isolation. This raises questions about potential impairments in social abilities, particularly in recognizing facial emotions, which may be linked to the subjective complaints of reduced quality of life in individuals with insomnia.

Several studies have explored facial emotion recognition in insomnia, with some indicating impairments in emotion recognition or evaluation of emotion intensity. Others demonstrated deficits in recognizing specific emotions (such as anger) or representations (such as fatigue), which were associated with attentional deficits and changes in visual fixation points in eye-tracking studies.

However, some authors found no significant association between insomnia complaints and impaired facial emotion recognition. Facial emotion recognition has been studied using eye-tracking in major depressive episodes, attention-deficit/hyperactivity disorder (ADHD), and autism spectrum disorders. Eye-tracking studies have revealed attentional biases toward negative emotions in depression and deficits in visual attention to the eye region in autism, contributing to impaired facial emotion recognition. To date, no study has compared facial emotion recognition abilities between individuals with insomnia and a control group, considering attentional deficits and emotional dysregulation described in insomnia.

Methods The study aims to compare two groups: one with isolated insomnia (without associated psychiatric disorders) and a control group (without insomnia or psychiatric disorders). Patients with psychiatric or addictive disorders will be excluded based on Diagnostic and Statistical Manual of Mental Disorders, version 5 (DSM-V) psychiatric interviews. Participants aged over 65 or under 18 will also be excluded to mitigate potential biases related to dementia and cognitive alterations not related to insomnia.

The insomnia group will consist of individuals seeking care at the Sleep Center of Angers University Hospital for chronic insomnia (lasting more than 3 months). Insomnia will be confirmed using the Insomnia Severity Index (ISI), with a score exceeding 15, while individuals with subclinical insomnia (ISI score between 7 and 15) will be excluded. The control group will have an ISI score below 7 (indicating the absence of insomnia).

The main objective is to determine whether facial emotion recognition differs between the insomnia and control groups. Secondary objectives include assessing differences between explicit facial emotion recognition tests (controlled conditions) and eye-tracking tests (implicit memory) in both groups to evaluate attentional biases. Additionally, the study aims to explore differences in facial emotion recognition tests based on emotional regulation profiles (adaptive or non-adaptive regulation).

Expected Results The hypothesis is that facial emotion recognition under controlled conditions (explicit memory) will not differ between the insomnia and control groups. However, differences are expected in implicit memory tests (eye-tracking) due to the attentional deficits previously described in insomnia. Additionally, variations in facial emotion recognition are anticipated based on emotional regulation profiles, which may influence facial emotion recognition in insomnia.

The study's findings could contribute to a better understanding of cognitive complaints related to insomnia, especially in the realm of social interactions, by objectively assessing and specifying potential biases. This research may also inform targeted therapeutic approaches, particularly in cognitive-behavioral therapy, focusing on cognitive remediation and restructuring. Ultimately, the study's outcomes could guide the development of specific rehabilitation programs centered on facial emotion recognition, emotional deficits, and emotional dysregulation in insomnia.

DETAILED DESCRIPTION:
Methods Each group will undergo two facial emotion recognition tests, one under controlled conditions with unlimited time (explicit memory recognition) and the other using eye-tracking to assess attentional biases (implicit memory recognition). The two groups will then be compared to determine differences in facial emotion recognition abilities between insomnia and control groups (primary outcome). The study will also explore the same abilities using eye-tracking (considering attentional deficits and visual fixation) and compare the results based on emotional regulation profiles (considering the potential impact of emotional dysregulation, which is more frequently described in insomnia).

Data will be collected by a physician using paper-based questionnaires and entered into an anonymized database on the hospital's restricted network drive. The anonymized participant code will consist of the first letter of the first name, first letter of the last name, group (0: controls/1: insomnia), and inclusion number (e.g., JG-0-001). This research project will be conducted in collaboration with the Adult Psychiatry Service, the Sleep Center, and the Ophthalmology Service at Angers University Hospital and will be part of the Laboratory of Psychology of the Pays de la Loire (LPPL - Research Unity 4638).

ELIGIBILITY:
Pre-inclusion criteria

* Age between 18 and 65
* Signed consent to participate in the study
* Person affiliated to or benefiting from a social security scheme
* For insomnia group: known insomnia (patient treated for insomnia)

Inclusion criteria:

* Insomnia group: ISI >14 (between 15 and 28 = clinical insomnia)
* Control group: ISI < 8 (between 0 and 7 = no insomnia)

Non-pre-inclusion criteria

* Known psychiatric disorders (Characterized depressive episode, Bipolar disorder, Schizophrenia and other delusional disorders, Specified anxiety disorder (social anxiety, generalized anxiety disorder), Obsessive-compulsive disorder (OCD), Eating disorders, Neurodevelopmental disorders (ASD, ADHD), Active addictive disorders (excluding tobacco), ...)
* Taking antidepressant, neuroleptic or thymoregulator medication
* Taking a benzodiazepine with a long half-life (>12 hours)
* Condition requiring hospitalization in the month preceding the study
* Known sequelae or progressive neurological disease
* Known significant ophthalmological condition
* Pregnancy or breast-feeding
* Person deprived of liberty by judicial or administrative decision
* Person subject to a legal protection measure
* Person under psychiatric care without consent
* For control group: no known insomnia

Non-inclusion criteria :

- Psychiatric disorders identified during psychiatric interview

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Facial emotion recognition test (TREF test) in insomnia and control | 10 minutes
  The error rate on facial recognition test (in percent)
Facial emotion recognition test (TREF test) in insomnia and control | 10 minutes
  The intensity of the emotion on facial recognition test (in percent)
Facial emotion recognition test (TREF test) in insomnia and control | 10 minutes
  Response time on facial recognition test (in second)

SECONDARY OUTCOMES:
Attentional bias | 10 minutes
  Measurement of errors rate on facial recognition test (TREF test) with eye-tracking dispositif (in percent)
Attentional bias | 10 minutes
  Intensity of the recognized emotion on facial recognition test in eye-tracking (in percent)
Attentional bias | 10 minutes
  Measurement of first fixation duration on facial recognition test in eye-tracking (in second)
Attentional bias | 10 minutes
  Measurement of duration of fixation on eyes (of face photography in the test) on facial recognition test in eye-tracking
Attentional bias | 10 minutes
  Measurement of duration of fixation on nose (of face photography in the test) on facial recognition test in eye-tracking
Attentional bias | 10 minutes
  Measurement of duration of fixation on mouth (of face photography in the test) on facial recognition test in eye-tracking
Emotional dysregulation bias | 5 minutes
  Cognitive Emotional Regulation Questionnaire (CERQ) test. The CERQ is made up of 36 assertions with multiple related propositions i.e. "almost never, sometimes, regularly, often, almost always" corresponding to a score between 1 and 5. It identifies two main types of emotional regulation strategy profile according to the scores obtained on the various questions, each ranging from 4 to 20 : measures adaptive regulation (sub-types: acceptance, positive centering, action centering, positive re-evaluation, perspective-taking) and non-adaptive regulation (sub-types: self-blame, rumination, catastrophism, blaming others).
  others).

IPD SHARING:
Plan to Share IPD: No